CLINICAL TRIAL: NCT03381716
Title: Correlation Between Sex and Prognosis of Acute Aortic Dissection in the Chinese Population
Status: Completed | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, Correlation between sex and prognosis of acute aortic dissection in the Chinese population, Shenyang Northern Hospital
Other Study IDs: SYNH-20171207
Record Dates: First submitted 2017-12-11; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Acute Aortic Dissection; Sex Role
Keywords: aortic dissection; sex; treatment
MeSH Terms: conditions — Aortic Dissection; Coitus | interventions — Pharmaceutical Preparations; Endovascular Aneurysm Repair; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male: Drug:Beta-blocker,Angiotensin II receptor blocker,Angiotensin-converting enzyme,Calcium-channel blocker,Aspirin,Statin
  Interventions: Drug: drug; Procedure: Surgery
- female: Drug:Beta-blocker,Angiotensin II receptor blocker,Angiotensin-converting enzyme,Calcium-channel blocker,Aspirin,Statin
  Interventions: Drug: drug; Procedure: Surgery

INTERVENTIONS:
Drug: drug — Application bracket
  Other Names: thoracic endovascular aortic repair
Procedure: Surgery — Surgery

SUMMARY:
The study evaluated the prevalence, presentation, management, and prognosis of coronary heart disease differ according to sex.

DETAILED DESCRIPTION:
The study included 884 patients enrolled in our institute between June 2002 and May 2016. Considering psychosocial factors, treatments, and the outcomes in men versus those in women with acute aortic dissection, explored the association of sex with psychosocial characteristics and mortality risk. Of 884 patients, 211 (23.9%) were women. The median duration of follow-up was 2.9 years (25th -75th percentiles: 1-4 years ).

ELIGIBILITY:
Inclusion Criteria:

* acute aortic dissection

Exclusion Criteria:

* Chronic aortic dissection

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 884 (Actual)
Dates: Start 2002-06-19 (Actual); Primary Completion 2016-05-29 (Actual); Study Completion 2016-05-29 (Actual)

PRIMARY OUTCOMES:
The outcome measure describes aortic disease-related death，aortic dissection, paraplegia, myocardial ischemia, renal insufficiency and other aortic complications. | 2.9years
  The study's primary endpoint during the follow up was the composite of aortic disease-related death, aortic dissection, paraplegia, myocardial ischemia, renal insufficiency and other aortic complications during follow-up.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bossone E, LaBounty TM, Eagle KA. Acute aortic syndromes: diagnosis and management, an update. Eur Heart J. 2018 Mar 1;39(9):739-749d. doi: 10.1093/eurheartj/ehx319. PMID 29106452